CLINICAL TRIAL: NCT02540733
Title: MRI Study of the Structural and Functional Rehabilitation in the Cerebral Infarction Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Minming Zhang, Chief,Department of Radiology,The 2nd Affiliated Hospital of Zhejiang University, School of Medicine, Zhejiang University
Other Study IDs: 81271530
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cerebral Stroke; Diabetes Mellitus
Keywords: cerebral infarction; diabetes; rehabilitation; MRI
MeSH Terms: conditions — Stroke; Diabetes Mellitus; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic stroke
- Non-diabetic storke

SUMMARY:
Diabetes mellitus (DM) plays an important role in the occurrence of the cerebral infarction (CI). Clinical studies have demonstrated that the CI patients with DM had a poor prognosis compared with those without DM. Previous magnetic resonance imaging (MRI) studies have shown that patients with DM had abnormalities in cerebral vessels, nerves and functions, similar with the findings in mice models. In this study, with multi-modal MRI technologies, investigators tend to observe structural and functional changes of the brain in both DM and non-DM CI patients and assess their neural rehabilitation using clinical scales in the following 6 months. Investigators also expect to find out dynamic changes of brain structure and function, to reveal the weights of factors including brain blood vessels, nerves and function remodeling related with stroke recovery, as well as the potential mechanism in CI patients with DM.

ELIGIBILITY:
Inclusion Criteria:

1. ﬁrst-ever ischemic stroke;
2. single infarct in the distribution of the middle cerebral artery;
3. no evidence of hemorrhagic infarction;
4. age greater than 18 years;
5. admission between 3 and 7 days after stroke onset;
6. National Institute of Health Stroke Score (NIHSS) score of 4 to 21 on admission and
7. no thrombolytic or recanalization therapies.

Exclusion Criteria:

1. atrial fibrillation;
2. history of neurological or psychiatric disorders;
3. pre-stroke modified Rankin scale (mRS) > 1;
4. life expectancy < 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: with a definition of stroke within 3 to 7 days after onset
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-01-01; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) | 6 months
  scores range from 0 (no symptoms) to 6 (dead)
National Institute of Health Stroke Score | 6 months
  scores ranging from 0 to 42 (the higher the score, the greater the function deficits)
Barthel index | 6 months
  score ranging from 0 (totally dependent) to 100 (completely independent)

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of Zhejiang University, School of Medicine,, Hangzhou, Zhejiang, China